CLINICAL TRIAL: NCT05953519
Title: Meeting an Unmet Need in Multiple Sclerosis (MS): An Evaluation of the Effectiveness of a Transdiagnostic Psychological Treatment and Its Outcomes
Brief Title: Meeting an Unmet Need in Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Lauren Strober, Principle Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1205-23
Record Dates: First submitted 2023-04-12; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor is blinded to the group assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol intervention (Experimental): The Unified Protocol consists of 12-weeks, virtual, group sessions focused on reducing depression and anxiety through: (1) Increasing emotional awareness; (2) Cognitive restructuring against dysfunctional beliefs; (3) Changing action tendencies associated with disordered emotions; (4) Preventing emotional avoidance and utilizing emotion exposure techniques; (5) Providing mutual help among group members; and (6) Providing opportunities for corrective experiences.
  Interventions: Behavioral: Unified Protocol
- Control group (No Intervention): The control group will not receive any intervention and will complete the same baseline and follow-up assessments.

INTERVENTIONS:
Behavioral: Unified Protocol — The Unified Protocol is a transdiagnostic intervention developed to treat depression and anxiety.
  Arms: Unified Protocol intervention

SUMMARY:
The primary objectives of this study is to examine the efficacy of the Unified Protocol in decreasing depression and anxiety among individuals with MS and the secondary outcomes (e.g., improved well-being, QOL, coping, etc.) that may occur in tandem.

DETAILED DESCRIPTION:
The primary objectives of this study is to examine the efficacy of the Unified Protocol in decreasing depression and anxiety among individuals with MS and the secondary outcomes (e.g., improved well-being, QOL, coping, etc.) that may occur in tandem.

To achieve this, the investigation has the following specific aims:

Specific Aim 1: Conduct a pilot Randomized Controlled Trial (RCT) of the Unified Protocol among individuals with MS to determine the effectiveness of the intervention in reducing depression and anxiety.

Hypothesis 1: Individuals who participate in the Unified Protocol intervention will report a decrease in their depression and anxiety compared to individuals in the control group.

Specific Aim 2: Conduct a pilot RCT of the Unified Protocol among individuals with MS to determine the effectiveness of the intervention in improving secondary outcomes of psychological well-being, QOL, coping, and MS symptomatology over time.

Hypothesis 2: Individuals who participate in the Unified Protocol intervention will report an increase in psychological well-being, QOL, coping, and MS symptomatology over time compared to participants in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis
* 18 years of age or older
* Experiencing significant depression and/or anxiety
* English-speaking
* Able to provide informed consent
* Access to the internet

Exclusion Criteria:

* History of any other neurological illness (e.g. traumatic brain injury, epilepsy, dementia)
* Current participation in another randomized controlled trial
* Cognitive impairment that would affect my ability to fully participate in the group
* Unable to attend group sessions
* Active participation in another formal clinical group or psychological therapy
* Any other medical or psychological condition that, in the judgement of the investigators, prevents successful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) - Change in Depression | Baseline, 12 weeks, 24 weeks
  Self-report measure of depression. Scores range from 0-21 with higher scores indicating greater depression.
Hospital Anxiety and Depression Scale (HADS) - Change in Anxiety | Baseline, 12 weeks, 24 weeks
  Self-report measure of anxiety. Scores range from 0-21 with higher scores indicating greater anxiety.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) - Change in Fatigue | Baseline, 12 weeks, 24 weeks
  Self-report measure of fatigue. Scores range from 0-84 with higher scores indicating greater fatigue.
Pittsburgh Sleep Quality Index (PQSI) - Change in Sleep | Baseline, 12 weeks, 24 weeks
  Self-report measure of sleep. Scores range from 0-21 with higher scores indicating greater sleep problems.
MOS Pain Effects Scale (PES) - Change in Pain | Baseline, 12 weeks, 24 weeks
  Self-report measure of pain. Scores range from 0-30 with higher scores indicating greater pain.
General Self-Efficacy Scale (GSES) - Change in Self-efficacy | Baseline, 12 weeks, 24 weeks
  Self-report measure of self-efficacy. Scores range from 10-40 with higher scores indicating greater self-efficacy.
University of Washington Self-Efficacy Scale - Change in MS specific self-efficacy | Baseline, 12 weeks, 24 weeks
  Self-report measure of disease self-efficacy. Scores range from 0-100 (T-scores) with higher scores indicating greater self-efficacy.
University of Washington Resilience Scale - Change in Resilience | Baseline, 12 weeks, 24 weeks
  Self-report measure of resilience. Scores range from 8-40 with higher scores indicating greater resilience.
COPE inventory - Change in Coping | Baseline, 12 weeks, 24 weeks
  Self-report measure of coping. Scores range from 4-16 for each coping scale with higher scores indicating greater coping.
Benefit Finding in Multiple Sclerosis (BFIMS) - Change in Benefit-finding | Baseline, 12 weeks, 24 weeks
  Self-report measure of positive coping. Scores range from 43-129 for the total scale with higher scores indicating greater benefit-finding.
Satisfaction with Life Scale (SWLS) - Changes in Quality of Life | Baseline, 12 weeks, 24 weeks
  Self-report measure of quality of life and satisfaction. Scores range from 5-35 with higher scores indicating greater life satisfaction.
Flourishing Scale (FS) - Change in Quality of Life | Baseline, 12 weeks, 24 weeks
  Self-report measure of quality of life. Scores range from 8-56 with higher scores indicating greater quality of life.
Ryff Psychological Well-being Scales (RYFFPWB) - Changes in well-being | Baseline, 12 weeks, 24 weeks
  Self-report measure of psychological well-being. Scores range from 14-84 for each subscale with higher scores indicating greater psychological well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided